CLINICAL TRIAL: NCT04915287
Title: Efficacy of Avatrombopag in Thrombocytopenic Patients With Chronic Liver Disease Undergoing an Elective Procedure: A Prospective Non-randomized Controlled Trial
Brief Title: Efficacy of Avatrombopag in Thrombocytopenic Patients With Chronic Liver Disease Undergoing an Elective Procedure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Chief physician, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2021-240-02
Record Dates: First submitted 2021-05-23; First posted 2021-06-07 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Thrombocytopenia; Drugs; Chronic Liver Disease
Keywords: Thrombocytopenia; Chronic Liver Disease; Avatrombopag; Invasive procedure
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag; Platelet Transfusion; Dosage Forms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Avatrombopag (Experimental): Oral administration of Avatrombopag Maleate Tablets to the thrombocytopenic patients with chronic liver disease undergoing an elective procedure whose mean baseline platelet count is less than 50 × 10^9/L. RhuTPO, rhIL-11, Romiplostim, Eltrombopag, or Lusutrombopag, etc., are prohibited during the trial.
  Interventions: Drug: Avatrombopag maleate
- Conventional treatment (Experimental): Conventional treatment (platelet transfusion if needed or rhuTPO, rhIL-11, Romiplostim, Eltrombopag, or Lusutrombopag, etc.) to the thrombocytopenic patients with chronic liver disease undergoing an elective procedure whoes mean baseline platelet count is less than 50 × 10^9/L.
  Interventions: Biological: Platelet transfusion; Drug: Medicine

INTERVENTIONS:
Drug: Avatrombopag maleate — 1. Mean baseline platelet count 40 to less than 50 × 10^9/L: 40mg Avatrombopag QD × 5 days from 10-13 days pre-procedure
  2. Mean baseline platelet count less than 40 × 10^9/L: 60mg Avatrombopag QD × 5 days from 10-13 days pre-procedure
  Other Names: Doptelet
  Arms: Avatrombopag
Biological: Platelet transfusion — Mean baseline platelet count less than 50 × 10^9/L pre-procedure: platelet transfusion if needed
  Arms: Conventional treatment
Drug: Medicine — Mean baseline platelet count less than 50 × 10^9/L pre-procedure: rhuTPO, rhIL-11, Romiplostim, Eltrombopag, or Lusutrombopag, etc.
  Other Names: Other drugs
  Arms: Conventional treatment

SUMMARY:
In this study, investigators aimed to evaluate the efficacy of Avatrombopag in thrombocytopenic patients with chronic liver disease undergoing an elective invasive procedure through a prospective, non-randomized controlled, multicenter clinical trial. The patients were non-randomly assigned to the Avatrombopag group (119 patients) and the conventional treatment group (357 patients). The primary endpoint was the proportion of patients not requiring prophylactic platelet transfusion or rescue therapy due to bleeding from grouping up to 10 days post-procedure. Second endpoints included the proportion of patients achieving a platelet count of ≥50x10^9/L and the mean change in platelet count from baseline at the time before the procedure, the proportion of patients requiring platelet transfusion and the mean platelet transfusion units per capita, the incidence of bleeding events (WHO≥2 and requiring rescue therapy), the imaging evaluations of bleeding events, the incidence of adverse events, the changes in life quality between two groups before and after treatment, and the pharmacoeconomic index of two groups.

Note: According to the results of interim statistical analysis (200-300 cases), it is up to the sponsor to decide whether to terminate the study in advance or increase the number of included cases at a later stage.

DETAILED DESCRIPTION:
Thrombocytopenia is a common complication of chronic liver disease (CLD), which severity increases with the aggravation of CLD. TPO, the primary physiological regulator of platelet production, is mainly produced by the liver. With the progressive liver injury in patients with CLD, TPO production decreases, resulting in the reduction of platelet production and thrombocytopenia, which cause the significantly increased risk of bleeding during the invasive procedure in these patients and pose a severe challenge to clinical management.

Platelet transfusion is a standard clinical treatment for CLD-related thrombocytopenia. Whether prophylactic platelet transfusion is needed before elective invasive procedure depends on the level of platelet count and the judgment of medical staff on the risk of bleeding in those procedures. Clinically, without effective preventive treatment in severe thrombocytopenia (PLT< 50×10^9/L), the risk of bleeding in related procedures is high, the hospitalization is prolonged after bleeding, and other post-procedure complications may occur. However, repeated prophylactic platelet transfusion may lead to ineffective platelet transfusion.

ADAPT-1 and ADAPT-2 were identical design randomized, double-blinded, placebo-controlled, international multicenter phase III clinical trials. They confirmed that 1. Avatrombopag could significantly increase the platelet count in patients with chronic liver disease with severe thrombocytopenia (PLT<50×10^9/L), thus reducing the proportion of platelet transfusion or rescue due to bleeding in adult patients with chronic liver disease-associated thrombocytopenia undergoing elective invasive procedures; 2. In terms of safety, the incidence of adverse events in the Avatrombopag group was comparable to that in the placebo group. At present, Avatrombopag has been successively approved in Europe, the United States, and China for adult patients with chronic liver disease-associated thrombocytopenia undergoing elective invasive procedures.

Avatrombopag is effective and safe in raising platelet count in patients with chronic liver disease. In addition, it has the characteristics of no risk of neutralizing antibody generation from small molecules and convenient oral administration.

The purpose of this study was to observe the clinical benefit of Avatrombopag to raise platelet count in adult patients with chronic liver disease-associated thrombocytopenia who received elective high-risk invasive procedures and to validate the efficacy and safety of Avatrombopag further in Chinese population with different spectrum of etiology in chronic liver disease.

Note: According to the results of interim statistical analysis (200-300 cases), it is up to the sponsor to decide whether to terminate the study in advance or increase the number of included cases at a later stage.

ELIGIBILITY:
Inclusion Criteria:

1. Both men and women are at least 18 years old at the time of signing the informed consent;
2. Baseline platelet count<50×10^9/L;
3. Patients with chronic liver disease undergo elective invasive procedures with high bleeding risk. The invasive procedures include liver/kidney biopsy or ablation, biliary drainage/stent implantation, cholecystostomy, transjugular intrahepatic portal venous shunt, nephrostomy and catheterization, chemotherapy embolization, abdominal/pelvic/retroperitoneal/mediastinal biopsy or ablation, endoscopic polypectomy, endoscopic stricture dilation or mucosal resection, balloon-assisted enteroscopy, percutaneous endoscopic gastrostomy, endoscopic retrograde cholangiopancreatography with sphincterotomy (ERCP + EST), endoscopic ultrasound with fine-needle aspiration (EUS-FNA), cyst gastrostomy, dental extraction, angiography or interventional venography and therapeutic coronary angiography such as PCI), and intraarticular injection, etc.;
4. Be able to understand the study and is willing to follow all study procedures, and voluntarily sign informed consent before screening;
5. According to the opinions of the researchers, it can meet the requirements of this study.

Exclusion Criteria:

1. Subjects with a history of arterial or venous thrombosis within six months before baseline;
2. Subjects with a known history of the hereditary prethrombotic syndrome include thrombin factor V Leiden mutation, prothrombin G20210A mutation, or hereditary antithrombin III (ATIII) deficiency;
3. Subjects could not suspend anticoagulants or antiplatelet therapy within one week preoperatively, such as heparin (within 24 hours before the procedure for Low molecular weight heparin), warfarin, rivaroxaban, dipyridamole, non-steroidal anti-inflammatory drugs, aspirin, verapamil, ticlopidine, clopidogrel, glycoprotein IIb/IIIa antagonists, and erythropoietin, etc.;
4. Subjects could not suspend Chinese patent medicines within three days before the procedure to promote blood circulation and remove blood stasis, such as pseudo-ginseng, red-rooted salvia, etc.;
5. Subjects received thrombopoietin receptor agonists within two weeks before enrolment, such as rhuTPO, Romiplostim, Eltrombopag, Avatrombopag, or Lusutrombopag, etc. Subjects received rhIL-11 within two weeks before enrolment. Moreover, subjects received platelet transfusion within one week before enrolment;
6. Subjects with thrombocytopenia caused by primary blood diseases (immune thrombocytopenia, myelodysplastic syndrome, etc.) or drugs (such as chemotherapy drugs, targeted therapy drugs, immune checkpoint inhibitors, etc.). Exceptions: Subjects are allowed to receive targeted drugs that do not cause thrombocytopenia, provided that these targeted therapy drugs are discontinued for a while to reduce the risk of bleeding, as follows: Bevacizumab for four weeks (6 weeks for patients with coagulation abnormality), lumvaritinib, sorafenib, pazopanib, axitinib, cabozantinib, anlotinib, apatinib, nidanib, and sunitinib for one week, and fuquanitinib for two weeks, etc.;
7. Subjects scheduled for splenic embolization (excluding those with persistent low platelet counts after splenic embolization or splenectomy);
8. Concomitant medical histories (e.g., gastrointestinal bleeding within three months; high risk of thrombosis, e.g., portal vein blood flow velocity < 10cm/s) may prevent subjects from completing the study safely;
9. Subjects are allergic to avatrombopag or any of its excipients;
10. A woman who is pregnant or who intends to become pregnant;
11. Subjects participate in another clinical study using any exploratory drug or device within 30 days before their baseline visit; Participation in observational studies is permitted;
12. The investigator considers that any accompanying medical history of the subject may affect the subject's ability to complete the study safely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2021-06-06 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients not requiring prophylactic platelet transfusion | From grouping up to 10 days post-procedure
  The proportion of patients not requiring prophylactic platelet transfusion
The proportion of patients not requiring rescue therapy due to bleeding | From grouping up to 10 days post-procedure
  The proportion of patients not requiring rescue therapy due to bleeding

SECONDARY OUTCOMES:
The proportion of patients achieving a platelet count of ≥50x10^9/L | The time before the procedure in the procedure day
  The proportion of patients achieving a platelet count of ≥50x10^9/L
The mean change in platelet count from baseline | The time before the procedure in the procedure day
  The mean change in platelet count from baseline
The proportion of patients requiring platelet transfusion | From grouping up to 10 days post-procedure
  The proportion of patients requiring platelet transfusion
The mean platelet transfusion units per capital | From grouping up to 10 days post-procedure
  The mean platelet transfusion units per capital
The incidence of bleeding events | From grouping up to 10 days post-procedure
  The recorded bleeding events included WHO≥2 and requiring rescue therapy
The imaging evaluations of bleeding events | From grouping up to 10 days post-procedure
  The imaging evaluations of bleeding events
The Incidence of adverse events | From grouping up to 10 days post-procedure
  The Incidence of adverse events
The changes in life quality between two groups assessed by EuroQol Five Dimensions Questionnaire | From grouping up to 10 days post-procedure
  The changes in life quality between two groups assessed by EuroQol Five Dimensions Questionnaire (EQ-5D) include mobility, self-care, usual activities, pain/discomfort, anxiety/depression. All five dimensions are described by three problem levels corresponding to patient response choices. The EQ-5D total score from the five dimensions ranges from 0 (worst health state) to 1 (perfect health state), and 1 reflects the best outcome.
The pharmacoeconomic indexes of two groups | From grouping up to 10 days post-procedure
  The pharmacoeconomic indexes include the cost of examination, the cost of medicine in platelet-raising, the cost of preventive measures for bleeding, the cost related to bleeding events, the cost of adverse events and the cost of health insurance, which are recorded in Chinese Yuan.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No